CLINICAL TRIAL: NCT01408069
Title: Multicentric, Randomizade, Double Blind, Double Dummy To Non-Inferiority Comparison Of Migrane® Versus Parcel ® For Treatment Of Tensional Cephaleia
Brief Title: Non-Inferiority Comparison of Migrane® Versus Parcel ® For Treatment of Tensional Cephaleia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study canceled by decision strategically.
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACHEMS0211
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Tensional-type Headache
Keywords: headache; migraine
MeSH Terms: conditions — Headache; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIGRANE (Experimental): 1 to 2 tablets ergotamine 1mg + caffeine 100mg + acetylsalicylic 350 mg + homatropine 1,2 mg
  Interventions: Drug: MIGRANE
- PARCEL (Active Comparator): 1 to 2 tablets(ergotamine 1mg + paracetamol 450 mg + caffeine 40 mg)
  Interventions: Drug: PARCEL

INTERVENTIONS:
Drug: MIGRANE — 1 to 2 tablets(ergotamine 1mg + caffeine 100mg + acetylsalicylic 350 mg + homatropine 1,2 mg)
  Arms: MIGRANE
Drug: PARCEL — 1 to 2 tablets(ergotamine 1mg + paracetamol 450 mg + caffeine 40 mg)
  Arms: PARCEL

SUMMARY:
The purpose of this study is to evaluate the non-inferiority clinical efficacy of two different associations of drugs in the treatment of patients diagnosed with tensional-type headache in accordance with International Headache Society guidelines.

DETAILED DESCRIPTION:
* Open-label, non-inferiority, prospective, parallel group, intent to treat trial.
* Experiment duration: 56 days.
* 04 visits (days -7, 0, 28 and 56).
* Efficacy will be evaluated for 10 episodes of tension-type headache.
* Adverse events evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the study procedures agree to participate and give written consent.
2. Tensional-type headache patients according to the International Headache Society criteria.
3. Corporal body indices < 40.

Exclusion Criteria:

1. Pregnancy or risk of pregnancy.
2. Lactation
3. Use of acetylsalicylic acid or corticosteroids or immunosuppressive therapy.
4. Use of immunosuppressive drugs.
5. Alterations of laboratory selective tests.
6. Drugs or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in relieve headache symptoms. | 1 hour
  The evaluation of efficacy will be determined based on comparison of the intensity of headache before and after 30, 60 and 90 minutes of initiation of treatment.

SECONDARY OUTCOMES:
Tolerability of study treatment | 56 days
  Tolerability will be assessed by the investigator through the number of adverse events definitely related to study medication. This relationship will be defined by applying the Naranjo algorithm.